CLINICAL TRIAL: NCT02924441
Title: A Study Attempting to Improve the Comfort During Screening Mammography
Brief Title: Women's Mammography Study to Improve Comfort During Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CTMS 16-0045; HSC20160392H (Other: University of Texas Health Science Center- San Antonio)
Record Dates: First submitted 2016-09-08; First posted 2016-10-05 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Pain
Keywords: Mammogram; Pain Management; Lidocaine
MeSH Terms: conditions — Pain; Agnosia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Right Breast Lidocaine and calming music (Experimental): Group 1 - right breast lidocaine & calming music
  Interventions: Other: Lidocaine; Other: Calming Music
- Right Breast Lidocaine and no music (Experimental): Group 2 - right breast lidocaine & no calming music
  Interventions: Other: Lidocaine; Other: No Music
- Left Breast Lidocaine and calming music (Experimental): Group 3 - left breast lidocaine & calming music
  Interventions: Other: Lidocaine; Other: Calming Music
- Left Breast Lidocaine and no music (Experimental): Group 4 - left breast lidocaine & no calming music
  Interventions: Other: Lidocaine; Other: No Music

INTERVENTIONS:
Other: Lidocaine — Applied to breast skin
  Other Names: Topicaine
Other: Calming Music — Played during mammography
  Arms: Left Breast Lidocaine and calming music; Right Breast Lidocaine and calming music
Other: No Music — No music played during mammography
  Arms: Left Breast Lidocaine and no music; Right Breast Lidocaine and no music

SUMMARY:
To determine in a randomized trial whether it is possible to decrease the discomfort and anxiety of mammography by using the local analgesic lidocaine, or by using calming music in patients receiving a mammogram.

DETAILED DESCRIPTION:
The study is designed to evaluate two methods of reducing pain and anxiety caused by mammography, one of the barriers to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Must either be getting her first mammogram or based on prior experience be expecting level 4 or 5 pain.
* Must have two breasts

Exclusion Criteria:

* May not have taken ibuprofen or other pain medication within the Space last 12 hours (ASA 81 mg dose is allowed).
* Must not have a contraindication for using lidocaine: e.g no history of allergic reactions to lidocaine.
* Must not have had history of breast cancer, breast surgery, radiation to the chest wall.
* Must not have broken or irritated skin (as determined by the study nurses).
* May not be lactating or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Questionnaire to determine the change (or difference) in pain level before and after mammogram | The questionnaires are completed before and after mammography, on the same day (questionnaire will be completed before leaving the mammography clinic the day of mammography).
  The questionnaires will be typically be completed about 60 minutes apart. The first questionnaire will be completed before any intervention. The second questionnaire will be administered at the earliest at about 35 minutes later (after application of the gels and performance of mammography). The longest interval between administration of the questionnaires would be 75 minutes (after which time the gel must be removed, per protocol).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kist, MD, Principal Investigator — CTRC @ UTHSCSA; Virginia Kaklamani, MD, Study Chair — CTRC @ UTHSCSA; Pamela Otto, MD, Study Chair — CTRC @ UTHSCSA
Locations (1):
- UT Health Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No